CLINICAL TRIAL: NCT05857397
Title: A Collaborative Trial of Niraparib to Evaluate Patients With Ovarian Cancer in the Expanded Access Program in Latin America
Acronym: CONOR
Status: Active, not recruiting | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: LACOG 1220
Record Dates: First submitted 2023-03-06; First posted 2023-05-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated within the EAPs with niraparib for ovarian cancer: This is an observational study; patients will not be exposed to clinical interventions different from those belonging to the standard of care.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — This is an observational study; patients will not be exposed to clinical interventions different from those belonging to the standard of care.

SUMMARY:
Data from niraparib treatment is not available in real-world setting in Latin America. The present study aims to collect data from patients treated with niraparib within the Latin America Expanded Access Program (EAP) in clinical practice in Brazil and Argentina and who meet the eligibility criteria for this study, without additional intervention.

DETAILED DESCRIPTION:
This is a multicenter, retrospective and prospective (bi-directional) patient chart review, observational (non-interventional) study, in the patients treated within the Latin America EAP. The study is planned to be conducted at oncology services distributed in Argentina and Brazil. Its multicenter nature aims to improve the representativeness of the study population in the region. Patient's medical records will be screened by local clinical staff to assess for eligibility according to selection criteria in the sites previously involved in the EAP. The follow-up data collection will be performed using a combination of medical records and patients' interviews. For patients that had interrupted the treatment before study start, the study comprises a single study visit with retrospective data collection from medical charts, followed by follow-up overall survival status, progression-free survival and time to next treatment performed by medical chart review or by phone call at month 12, month 24 and month 36 from the first dose of niraparib. For those that were still in treatment, data collection will be performed during the regular visits to the services involved in the study, using a combination of medical records abstraction and patient's interviews.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced OC in response following first line platinum-based chemotherapy who were treated with niraparib within the EAP in Argentina and Brazil;
* Patients who have received at least one dose of niraparib in the EAP.

Exclusion Criteria:

* Patients without medical record available (lost, empty or irretrievable clinical information).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients with diagnosis of advanced high-grade ovarian, fallopian tube or primary peritoneal cancer who are in response (complete or partial) following completion of first-line platinum-based chemotherapy, treated within the niraparib EAP.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety profile | through study completion, an average of 36 months
  To evaluate the safety profile, including dose modifications, of niraparib in patients with advanced ovarian cancer in response following first-line platinum-based chemotherapy treated in a real-world setting within the EAP.

CONTACTS AND LOCATIONS:
Overall Officials: Angélica Nogueira Rodrigues, Principal Investigator — Latin American Cooperative Oncology Group
Locations (16):
- Argentina (3):
  - COIP - Centro Oncologico Integral Pampeano, Santa Rosa, La Pampa Province
  - Sanatorio de la Mujer, Rosario, Santa Fe Province
  - Fundacion Medica de Rio Negro y Neuquen, Neuquén
- Brazil (13):
  - CINPAM - Centro Integrado de Pesquisa da Amazônia, Manaus, Amazonas
  - Hospital Santa Rita de Cássia, Vitória, Espírito Santo
  - NOB - Núcleo de Oncologia da Bahia (Oncoclínicas), Salvador, Estado de Bahia
  - Oncocentro de Minas Gerais (Oncoclínicas), Belo Horizonte, Minas Gerais
  - IOP Pesquisa - Instituto de Oncologia do Paraná, Curitiba, Paraná
  - HMV - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - CPO - Centro de Pesquisa em Oncologia do Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor de Barretos, Barretos, São Paulo
  - Hospital Amaral Carvalho de Jaú, Jaú, São Paulo
  - ICESP - Instituto do Câncer do Estado de São Paulo, São Paulo
  - BP - A Beneficência Portuguesa de São Paulo, São Paulo
  - Instituto D'Or de Pesquisa e Ensino SP, São Paulo
  - Pérola Byington Centro de Pesquisa, São Paulo

IPD SHARING:
Plan to Share IPD: No